CLINICAL TRIAL: NCT02970656
Title: A Pilot Study of Biomarkers of Stress in Youth Who Use Teens.Connect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Miller Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1503015414
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teens.Connect (Experimental): The Teens-Connect internet-based program has two complementary components - TEENCOPE and Managing Diabetes. Managing Diabetes consists of 5 sessions on educational content related to diabetes self management targeted to adolescents. TEENCOPE consists of a series of 5 sessions designed to increase children's sense of competence and mastery by retraining inappropriate or non-constructive coping styles and forming more positive styles and patterns of behavior. Each week a new 30-45 minute session is uploaded to a password-protected website on the Yale server for youth to complete. Youth are grouped with 8-12 peers who complete the same weekly sessions in an asynchronous manner. Youth interact with each other on an online discussion board moderated by a clinical psychologist.
  Interventions: Behavioral: Teens.Connect
- Control (No Intervention): Wait listing will serve as the control condition. Usual care at the Yale Pediatric Diabetes Center consists of quarterly visits with physicians and nurse practitioners, accessibility to nutritional and psychological consultation, and 24/7 on call service. Following completion of the 6 month data point, youth will be offered the opportunity to participate in the internet program.

INTERVENTIONS:
Behavioral: Teens.Connect — Teens.Connect combines two internet psycho-educational programs, TEENCOPE™, an internet version of coping skills training using a graphic novel format combined with social media, and an internet diabetes problem-solving educational program (Managing Diabetes)
  Arms: Teens.Connect

SUMMARY:
This feasibility/pilot study has three purposes. First, the investigators will determine the feasibility of collecting saliva to measure stress biomarkers over three days at home in youth. Second, the investigators will conduct a pilot study of the Teens.Connect Internet program for youth with type 1 diabetes to determine whether changes in stress biomarkers associate with self-reported perceived stress and HbA1c. Third, the investigators will examine the gene-environment interaction of the top 14 targeted candidate genes and epi-genome wide effects of teens' stress biomarkers and its influence on blood glucose levels over time.

DETAILED DESCRIPTION:
Intensive management of type 1 diabetes (T1D) among youth as recommended by the American Diabetes Association requires a complex set of self-management activities that create high levels of perceived stress in youth and families. In individuals exposed to chronic stress, such as that of a chronic condition, the body responds with physiological and hormonal responses to adapt. These responses can be harmful (e.g., higher glucose levels, higher HbA1c). Such harmful effects may be ameliorated by programs that reduce psychosocial stress.

The investigators have found an Internet-delivered coping skills training program combined with a diabetes education program significantly improved HbA1c and QOL for youth with T1D. Self-reported perceived stress mediated these outcomes. There has been little to no examination, however, of whether a reduction in self-reported perceived stress is associated with a reduction in biochemical markers of stress which could explain the positive impact on HbA1c. It is critically important to understand the physiologic as well as the psychosocial mechanisms associated with such interventions in order to improve glycemic control in youth with this chronic autoimmune condition. If such interventions affect biomarkers of stress, it would be important to strengthen the stress reduction activities embedded in such interventions, such as meditation, to further improve metabolic control. Thus, aims of this pilot/feasibility study are to:

1. Determine the feasibility and reliability of collection of saliva for the measurement of three stress biomarkers at awakening and 30-45 minutes later over 3 days at home in 20 youth (age 11-14 years). These biomarkers include cortisol to assess hypothalamic-pituitary-adrenal axis functioning; alpha-amylase (s-AA) to assess the sympathetic-adrenal-medullary system, and salivary immunoglobulin A (s-IgA) to assess stress-related immune changes. This aim will allow the investigators to determine the feasibility of recruiting youth to provide such data in a larger trial by assessing the percent of youth who agree to participate and adhere to the salivary collection protocol, using actigraphy to document awakening time and Medication Event Monitoring System (MEMS) caps monitoring to determine time of salivary collection. Patterns and variability of stress biomarker levels over 3 days will be used to assess intra-individual variability and relationships with self-reported daily stressors and self-reported perceived stress.
2. Conduct a pilot study of Teens.Connect, a combination of the investigators' previous TEENCOPE™ and Managing Diabetes programs with 40 youth to determine whether alterations in stress biomarkers are associated with self-reported perceived stress and HbA1c.
3. Assess epigenetic components of these responses by examining the gene-environment interaction of the top 14 targeted candidate genes and epigenome wide effects of teens' stress biomarkers and their influence on HbA1c levels over time. Candidate genes will be measured at baseline and DNA methylation patterns will be measured at baseline and then again at 6 months follow-up using the Oragene saliva collection kits.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with T1D for at least 6 months;
* age 11 to 14 years
* naïve to TEENCOPE and/or Managing Diabetes
* assent and parent/guardian consent to participate in the study

Exclusion Criteria:

* medical condition that impacts cortisol functioning
* takes medications that impact cortisol, except diabetes medications
* sleeps less than 6 hours per night
* smokes
* takes oral contraceptives

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Glycosylated Hemoglobin (HbA1c) | baseline
  Bayer Diagnostics DCA2000® (normal range = 4.2-6.3%)
Glycosylated Hemoglobin (HbA1c) | 6 months
  Bayer Diagnostics DCA2000® (normal range = 4.2-6.3%)

SECONDARY OUTCOMES:
Perceived Stress Scale | baseline
  A 14-item scale that measures the degree to which situations in one's life are appraised as stressful. Items assess feelings of stress, hassles, and coping during the past month. Respondents rate items on a 5-point Likert scale ranging from 0 (never) to 4 (very often), with higher scores indicative of greater perceived stress and less effective coping.
Perceived Stress Scale | 6 months
  A 14-item scale that measures the degree to which situations in one's life are appraised as stressful. Items assess feelings of stress, hassles, and coping during the past month. Respondents rate items on a 5-point Likert scale ranging from 0 (never) to 4 (very often), with higher scores indicative of greater perceived stress and less effective coping.
Adolescent Stress Questionnaire (ASQ) | baseline
  A 94-item inventory of common adolescent stressors. Each item (stressor) is rated on a 5-point Likert scale where 1=Not at all stressful (or is irrelevant to me); 2=A little stressful; 3=Moderately stressful; 4=Quite stressful; and 5=Very stressful.
Adolescent Stress Questionnaire (ASQ) | 6 months
  A 94-item inventory of common adolescent stressors. Each item (stressor) is rated on a 5-point Likert scale where 1=Not at all stressful (or is irrelevant to me); 2=A little stressful; 3=Moderately stressful; 4=Quite stressful; and 5=Very stressful.
Responses to Stress Questionnaire for Diabetes (RSQ) | baseline
  A 69-item scale asking the participant to report frequency of diabetes related stressors (12 items) and their responses to those stressors (57 items). Frequencies are reported on a 4-point scale ranging from 0 (never) to 3 (almost every day) for stressors, and 1 (not at all) to 4 (a lot) for stress responses.
Responses to Stress Questionnaire for Diabetes (RSQ) | 6 months
  A 69-item scale asking the participant to report frequency of diabetes related stressors (12 items) and their responses to those stressors (57 items). Frequencies are reported on a 4-point scale ranging from 0 (never) to 3 (almost every day) for stressors, and 1 (not at all) to 4 (a lot) for stress responses.
Stress Biomarkers | over 3 days at baseline
  cortisol, alpha-amylase (s-AA), and salivary immunoglobulin A (s-IgA) determined by salivary collection at awakening and 30-45 minutes later over 3 days
Stress Biomarkers | over 2 days at 6 months
  cortisol, alpha-amylase (s-AA), and salivary immunoglobulin A (s-IgA) determined by salivary collection at awakening and 30-45 minutes later over 2 days
Awakening and sleep time | over 3 days at baseline
  wrist-worn accelerometer
Awakening and sleep time | over 2 days at 6 months
  wrist-worn accelerometer
Genotype & DNA Methylation | baseline
  Saliva collection
DNA Methylation | 6 months
  Saliva collection

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Grey, DrPH, RN, Principal Investigator — Yale School of Nursing; Jacquelyn Taylor, PhD, PNP-BC, Principal Investigator — Yale School of Nursing
Locations (1):
- Yale School of Nursing, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No